CLINICAL TRIAL: NCT06077877
Title: A Phase 1/2 First-Time-in-Human, Open-label, Multicenter, Dose Escalation and Expansion Study of the Oral DNA Polymerase Theta Inhibitor (POLQi) GSK4524101 and the PARP Inhibitor (PARPi) Niraparib in Adult Participants With Solid Tumors
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics (PK), and Preliminary Anticancer Activity of GSK4524101 Alone or With Niraparib in Participants With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 219590
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
Keywords: POLQi; Niraparib; GSK4524101
MeSH Terms: conditions — Neoplasms | interventions — niraparib

STUDY DESIGN:
Masking Description: This is an open-label non-blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 - GSK4524101 Monotherapy (Experimental)
  Interventions: Drug: GSK4524101
- Part 1 - GSK4524101 plus Niraparib (Experimental)
  Interventions: Drug: GSK4524101; Drug: Niraparib
- Part 1 - GSK4524101 Food Effect Cohort (Experimental)
  Interventions: Drug: GSK4524101
- Part 2 - GSK4524101 plus Niraparib (Experimental)
  Interventions: Drug: GSK4524101; Drug: Niraparib
- Part 2 - Niraparib (Active Comparator)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: GSK4524101 — GSK452101 will be administered.
  Arms: Part 1 - GSK4524101 Food Effect Cohort; Part 1 - GSK4524101 Monotherapy; Part 1 - GSK4524101 plus Niraparib; Part 2 - GSK4524101 plus Niraparib
Drug: Niraparib — Niraparib will be administered.
  Arms: Part 1 - GSK4524101 plus Niraparib; Part 2 - GSK4524101 plus Niraparib; Part 2 - Niraparib

SUMMARY:
The primary purpose of this study is to determine the maximum tolerated dose of GSK4524101 monotherapy (MTD) and GSK4524101 in combination with niraparib (MTDc). The study consists of two parts - Part 1 (Dose Escalation) and Part 2 (Dose Expansion).

ELIGIBILITY:
Inclusion Criteria:

* More than or equal to (≥)18 years of age
* Eastern cooperative oncology group (ECOG) class 0-2
* Life expectancy of a minimum of 3 month
* Participant has histologically diagnosed advanced or metastatic solid tumor and has exhausted all standard of care treatment options (Part 1).
* Participant has metastatic, gBRCAmut, HER2-negative or HER2-low breast cancer who has completed at most 3 or more prior lines of therapy (Part 2).

Exclusion Criteria:

* Participant has not recovered (i.e., to Grade less than or equal to [≤1] or to baseline) from prior chemotherapy-induced AEs.
* Participant is currently participating in a treatment study or has participated in a study of any investigational agent within 4 weeks of the first dose of treatment.
* Participant has symptomatic uncontrolled brain or leptomeningeal metastases.
* Participant has a known additional malignancy that progressed or required active treatment within the last 2 years
* Participant has a known history of Myelodysplastic syndrome (MDS) or Acute myeloid leukemia (AML).
* Participant has uncontrolled hypertension with sustained systolic blood pressure (BP) >140 millimetres of mercury (mmHg) or diastolic BP >90 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Proportion of Participants with Dose Limiting Toxicities (DLTs) during DLT Observation Period | Up to 28 days
Part 1 - Proportion of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) based on Severity during DLT Observation Period | Up to 28 days
Part 1 - Duration of Treatment Emergent AEs and SAEs (Days) during DLT Observation Period | Up to 28 days
Part 1 - Percentage of Participants who receive all Planned Doses during DLT Observation Period | Up to 28 days
Part 1 -Percentage of Participants who require dosage interruptions, dose reductions, and drug discontinuations due to adverse reactions during DLT Observation Period | Up to 28 days
Part 2 - Confirmed Objective Response Rate (ORR) | Up to approximately 52 weeks
  ORR is the percentage of participants with an Investigator-assessed confirmed complete response and confirmed partial response to treatment, as assessed by Response Evaluation Criteria in Solid Tumor (RECIST) v1.1

SECONDARY OUTCOMES:
Part 1 - Area Under Curve (AUC) of GSK4364973 (Metabolite of GSK4524101) | Up to 21 weeks
Part 1 -Maximum Concentration (Cmax) of GSK4364973 (Metabolite of GSK4524101) | Up to 21 weeks
Part 1 - Time to Maximum Concentration of GSK4364973 (Metabolite of GSK4524101) | Up to 21 weeks
Part 1 - Half-life of GSK4364973 (Metabolite of GSK4524101) (Days) | Up to 21 weeks
Part 1 -Plasma Concentration of Niraparib | Up to 21 weeks
Part 1 - Number of Participants with TEAEs and SAEs based on Severity beyond DLT Observation Period | Up to approximately 24 weeks
Part 1 - Duration of TEAEs and SAEs (Days) beyond DLT Observation Period | Up to approximately 24 weeks
Part 2 - Number of Participants with TEAEs and SAEs based on Severity | Up to approximately 52 weeks
Part 2 - Duration of Treatment Emergent AEs and SAEs (Days) | Up to approximately 52 weeks
Part 2 - Progression-free Survival (PFS) | Up to approximately 52 weeks
  PFS is time from randomization to progressive disease or death from any cause, whichever is earlier, as assessed via RECIST v1.1 by Investigator assessment
Part 2 - Duration of Response (DOR) | Up to approximately 52 weeks
  DOR is defined as time from first documented PR or better to disease progression (as assessed by RECIST v1.1 by investigator assessment) or death whichever is earlier for participants who have achieved a CR or PR
Part 2 -Maximum Concentration (Cmax) of GSK4364973 (Metabolite of GSK4524101) | Up to 21 weeks
Part 2 - Minimum Concentration (Cmin) of GSK4364973 (Metabolite of GSK4524101) | Up to 21 weeks
Part 2 -Plasma Concentration of Niraparib | Up to 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (6):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Fairfax, Virginia
- Brazil (2):
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Vitória
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Panama (2):
  - GSK Investigational Site, Panama City
  - GSK Investigational Site, Punta Pacifica Panama City Panama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/